CLINICAL TRIAL: NCT03316781
Title: A Randomized, Double-Blind, Multi-Center, Active-Controlled, Parallel-Group Phase III Clinical Study to Compare the Efficacy and Safety of Recombinant Anti-TNFα Human Monoclonal Antibody Injection (HLX03) and Adalimumab Injection (Humira®) in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Study of Efficacy and Safety of HLX03 in Subjects With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX03-Ps03
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HLX03 group (Experimental)
  Interventions: Drug: HLX03
- adalimumab group (Active Comparator)
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: HLX03 — 80 mg SC at Week 0, 40 mg SC at Week 1, and 40 mg every other week thereafter.
  Arms: HLX03 group
Drug: adalimumab — 80 mg SC at Week 0, 40 mg SC at Week 1, and 40 mg every other week thereafter.
  Arms: adalimumab group

SUMMARY:
This is a multicenter, randomized, double-blind, positive drug parallel-group controlled clinical study in China to evaluate efficacy, safety, tolerability and immunogenicity of HLX03 and adalimumab (Humira) in subjects with moderate to severe plaque psoriasis. This study will recruit 216 subjects (18-75 years old, male and female) with moderate to severe plaque psoriasis. The 216 subjects will be randomly assigned per 1:1 ratio into the following two treatment groups (HLX03 OR Adalimumab). The study will be conducted in three periods, including the screening period, treatment period and follow-up period. For each participating subjects, the maximal length of the study will be 56 weeks (including up to four weeks of screening time).

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent.
2. Men or women is ≥18 and ≤ 75 years of age at time of screening.
3. Stable moderate to severe plaque psoriasis for at least 6 months before Screening.
4. Moderate to severe psoriasis as defined at Baseline by:

   BSA of ≥ 10% involvement at the Baseline visit. PGA score of ≥ 3 at the Baseline visit. PASI score of ≥ 12 at the Baseline visit.
5. Acceptable to systemic therapy, as judged by the investigator.
6. Previously received at least one traditional psoriasis treatment (for example, methotrexate, cyclosporine A, psoralen plus UVA or UVB, tretinoin, Chinese medicine, etc.), and was insensitive, intolerant, contraindicated to, or failed the treatment, as judged by the investigator.
7. At time of screening, lab tests have to meet the following:

   1. Hemoglobin ≥ 90 g/L
   2. WBC ≥ 3.5 × 10^9/L
   3. Platelets ≥ 100 × 10^9/L
   4. Serum creatinine ≤1.5 × upper limit of normal (ULN)
   5. AST and ALT ≤2 × ULN
8. For women of child-bearing age, a negative serum pregnancy test during screening, and a negative urine pregnancy test at baseline.
9. During the study to 150 days after the last dose of study medicine, subjects should use effective contraceptive measures
10. Subject is willing and able to comply with the visit schedule and other requirements of the study.

Exclusion Criteria:

1. At screening visit, subjects with erythrodermic psoriasis, pustule psoriasis, bit type psoriasis, drug-induced psoriasis, other skin lesions (such as eczema), other systemic autoimmune inflammatory lesions, which may affect the efficacy evaluation of the treatment.
2. The subject has surgery plan during the study period (excluding surgery that is related to the study disease), except that there will be no increased risk for the subjects or no influence on the study treatment or adherence to the study as judged by the investigator.
3. Participants were given the following treatment, or will be required to receive the following treatment during the study period:

   1. The use of topical drugs within the first two weeks before screening;
   2. The use of UVA and/or UVB treatment, and non-biological drugs (such as methotrexate, cyclosporin, tretinoin, traditional Chinese medicine, proprietary Chinese medicine, etc) within the first four weeks before screening;
   3. In the first 4 weeks before screening, the use of Etanercept or Etanercept; in the first 12 weeks before screening, the use of other biological agents
4. Subjects had live vaccination in the first four weeks before screening, or have the intention to receive live vaccination during the study period.
5. Subjects with history of mycobacterium tuberculosis infection, or with active tuberculosis, or with latent tuberculosis, or with suspected tuberculosis infection judged by clinical phenotypes.
6. Anti-HIV antibody positive, or antibody positive for treponema pallidum, or anti-HCV antibody positive, or HBV HBsAg and/or HBcAb positive at screening.
7. Accompanying active infection or history:

   1. Within 4 weeks before screening, systemic anti-infection treatment;
   2. Within 8 weeks before screening, severe infection with hospitalization or intravenous anti-infection treatment;
   3. Recurrent, chronic, or other active infections, which may increase the study risk as evaluated by the investigator.
8. Known malignancy or history of malignancy (except for the following: in situ skin squamous carcinoma after thorough treatment with no sign of recurrence, basal cell carcinoma, cervical cancer in situ, or skin squamous carcinoma at least five years prior to randomization with no signs of recurrence after treatment).
9. Ongoing, severe, progressive, or uncontrolled diseases, including but not limited to diseases at the endocrine system, blood system, urinary system, liver and gallbladder, respiratory system, nervous system, cardiovascular system, gastrointestinal system or infectious diseases, with increased risk to participate the study as assessed by the investigator.
10. The subjects with active neuropathies, such as multiple sclerosis, Guillain-Barre Syndrome, optic neuritis, transverse myelitis, or neurological symptoms suggestive of the demyelinating diseases of the central nervous system.
11. Moderate to severe heart failure (NYHA III/IV)
12. History of allergic reactions to the active components of the study drugs (HLX03 and adalimumab (Humira®)) and their formulation gradients, or medicines belonging to the same pharmacology and biological category.
13. Participated in another study and received an experimental related drugs within the previous 3 months before screening.
14. Pregnant or lactating women.
15. History of alcohol or substance abuse or dependence, mental disorders.
16. Any condition that will lead to no treatment benefit or affect efficacy evaluation, as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
Percentage improvement of PASI from baseline to Week 16 | Week 16
  Percent improvement of PASI from baseline to Week 16 will be calculated as the following formula: (PASI baseline-PASI Week 16) x 100% /PASI baseline

SECONDARY OUTCOMES:
PASI 75 response | Week 4, 8, 12, 16, 24, 32, 50
  75% or greater improvement in PASI score
PASI percent improvement | Week 4, 8, 12, 24, 32, 50
Static Physician's Global Assessment (sPGA) responses (with 0 or 1 being a positive result) | Week 4, 8, 12, 16, 24, 32, 50
Change of DLQI from baseline | Week 4, 8, 12, 16, 24, 32, 50

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, M.D., Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

REFERENCES:
- [Background] Cai L, Li L, Cheng H, Ding Y, Biao Z, Zhang S, Geng S, Liu Q, Fang H, Song Z, Lu Y, Li S, Guo Q, Tao J, He L, Gu J, Yang Q, Han X, Gao X, Deng D, Li S, Wang Q, Zhu J, Zhang J. Efficacy and Safety of HLX03, an Adalimumab Biosimilar, in Patients with Moderate-to-Severe Plaque Psoriasis: A Randomized, Double-Blind, Phase III Study. Adv Ther. 2022 Jan;39(1):583-597. doi: 10.1007/s12325-021-01899-0. Epub 2021 Nov 23. PMID 34816373